CLINICAL TRIAL: NCT01049178
Title: Antioxidant Enzyme Induction as a New Approach to Therapy in Patients With Asthma
Brief Title: Randomized Controlled Trial of Silymarin in Asthma
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Tina Hartert, Associate Professor of Medicine, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 090053
Record Dates: First submitted 2009-05-04; First posted 2010-01-14 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Atopic Asthma
Keywords: antioxidant enzymes; asthma; silymarin; RCT
MeSH Terms: conditions — Asthma | interventions — Silymarin; milk-thistle extract

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral silymarin dose (Experimental): Dose escalation study
  Interventions: Drug: Oral Silymarin; Drug: Oral Silymarin, maintenance dose
- placebo (Placebo Comparator): A randomized, double-masked, placebo-controlled cross-over clinical pilot investigation of an inducer of endogenous antioxidant enzymes, silymarin, in humans with atopic asthma.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral Silymarin — Dose Level 1: 1 capsules (1 cap at 140mg/cap) given three times per day for a total daily dose of 420 mg 28-days post Dose Level 1 Dose Level 2: 3 capsules (3 caps at 140mg/cap = 420 mg) given three times per day for a total daily dose of 1260 mg Day 56 (28-days post Dose Level 2) Dose Level 3: 5 capsules (5 caps at 140mg/cap = 700 mg) given three times per day for a total daily dose of 2100 mg Day 84 (28-days post Dose Level 3) We will evaluate change from baseline at each dose to determine the minimum effective dose.
  Other Names: Legalon; Milk Thistle
  Arms: Oral silymarin dose
Drug: Oral Silymarin, maintenance dose — The maintenance Silymarin dose will be selected based on the dose escalation study and will be dosed PO three times daily as recommended. Silymarin will be provided as a capsule S. marianum (70-80% silymarin), along with an identical appearance placebo capsule created by our investigational pharmacyAt each visit a questionnaire regarding daily symptoms and disease control, the asthma control test (ACT) will be completed, eNO measured, urine collected, spirometry (lung function) measured, venipuncture performed for blood collection (20 mL), as well as assessment of acceptability, toxicity, and masking.
  Other Names: Legalon; Milk Thistle
  Arms: Oral silymarin dose
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if intake of the antioxidant enzyme inducer, silymarin, will improve lung function and symptom scores in participants with asthma.

DETAILED DESCRIPTION:
SPECIFIC AIMS

Dietary intake of exogenous antioxidants has been shown to have only a modest impact on asthma inception and control. Our work has demonstrated that endogenous antioxidant enzyme concentrations are a far stronger predictor of asthma inception compared with dietary antioxidant intake and/or serum antioxidant concentrations. This is likely because we regulate oxidative stress to a greater extent, not by exogenous intake, but by antioxidant enzymes. The milk thistle plant extract, silymarin, has been shown to be an inducer of the endogenous antioxidant enzymes, superoxide dismutase and catalase. As reactive oxygen species have been implicated in the pathogenesis of asthma and, in atopic asthmatics, endogenous superoxide dismutase (SOD) enzyme levels are known to decrease, this supports that increasing SOD levels, either by induction of endogenous SOD or replacing a failed endogenous SOD enzyme system with a mimetic of the endogenous enzyme, would be beneficial and protective. We hypothesize that administration of silymarin, an inducer of antioxidant enzymes, to subjects with atopic asthma will increase antioxidant enzyme concentrations, decrease markers of oxidative stress, decrease indirect measures of airway inflammation that have been correlated with clinical outcomes (exhaled nitric oxide, eNO), and thus improve lung function and symptom scores in participants with asthma. To test this hypothesis we will conduct a randomized, double-masked, placebo-controlled cross-over pilot investigation of an inducer of endogenous antioxidant enzymes, silymarin, in asthma. No clinical trial has tested either silymarin, or any inducer of antioxidant enzymes in patients with asthma. We therefore aim to determine whether this novel treatment is effective, and if both inflammatory and clinical endpoints are improved with treatment.

Specific questions related to modification of endogenous antioxidant enzymes in prevalent asthma that this investigation aims to address are whether induction of antioxidant enzymes can alter inflammatory markers in asthma that are known to be linked with clinical endpoints, lung function and oxidant stress. Measurements of antioxidant enzymes will be made in blood samples prior to and following administration of silymarin; measures of systemic oxidative stress will be made in urine samples using an assay for isoprostanes, considered the most accurate marker of oxidative stress currently available; measures of airway inflammation will be measured using exhaled NO, and lung function testing and symptom control will be assessed as clinical measures of disease control.

Aim #1: To confirm that oral administration of silymarin in subjects with atopic asthma increases endogenous antioxidant enzymes. We hypothesize that silymarin will increase levels of antioxidant enzymes, superoxide dismutase activity, catalase activity, and glutathione peroxidase activity in subjects with atopic asthma. To test this hypothesis, we will first conduct a dose escalation study to determine optimal dosing, dose effect, and washout on airway inflammation, followed by a randomized, double-masked, placebo-controlled cross-over pilot investigation of supplementation with silymarin in subjects with atopic asthma with measurements of antioxidant enzyme activity pre-, during and at the completion of both active supplementation and placebo arms of the study.

Aim #2: To determine whether oral administration of silymarin to subjects with atopic asthma alters indirect measures of airway inflammation and systemic oxidative stress. We hypothesize that silymarin will decrease airway inflammation and measures of systemic oxidative stress. To test this we will assess indirect measures of airway inflammation, including exhaled nitric oxide and nitric oxide related products, and measures of systemic oxidant stress, urinary isoprostanes pre-, during and at the end of supplementation in the study subjects enrolled in this clinical trial.

Aim #3: To determine whether oral administration of silymarin to subjects with atopic asthma improves asthma morbidity, daily symptoms, disease control, disease exacerbations, and spirometry. We hypothesize that silymarin will improve asthma control and decrease morbidity. Although not powered for these outcomes, to test this hypothesis we will assess and evaluate the trends and magnitude of the effect of silymarin on asthma control, spirometry and disease exacerbations in the above study subjects.

Aim #4: To determine feasibility, acceptance of randomization, adherence to therapy, acceptance of drug delivery and dosing, ability to maintain blinding, and clinical effect size. The intent of this aim is to optimize the overall protocol design and procedures for a future larger study.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria Male or female subject with confirmed asthma, AND
* Age ≥ 18 years
* Asthma Control Test (ACT) Score of 15-20, AND
* Documented atopy by prick skin testing (most study participants will likely have participated in one of the investigators prior observational studies and will have had skin testing, if not, this will be performed at an in-person screening visit), AND
* For women: Not pregnant, as determined by a negative urinary pregnancy test at the initial visit(visit 1), AND at the start of the cross-over period (visit 4), AND using birth control

Exclusion Criteria:

* Known allergies to plants in the Asteraceae family (thistles, daisies, artichokes, kiwi)
* Non-asthmatic, or inadequate documentation which includes lack of signs and symptoms of asthma, or lack of prior confirmatory testing
* Pregnant
* Age < 18 years
* Non-English speaking
* Current smoker (current, or within last year)
* Chronic Obstructive Pulmonary Disease(COPD)
* Unable to swallow capsules
* Unable to obtain informed consent
* Unable to comply with avoidance of honey and propolis containing foods (which interfere with the silybin assays for measurement of plasma concentrations)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Exhaled nitric oxide (eNO), an indirect measure of airway inflammation that correlates with clinical asthma measures. | 20-40 weeks

SECONDARY OUTCOMES:
Spirometry, disease control, urinary isoprostanes, antioxidant enzyme concentrations, silybin concentrations, acceptability, ability to maintain blinding, effect size for secondary clinical outcomes. | 20-40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tina V. Hartert, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Wu P, Roberts LJ 2nd, Shintani AK, Sheller JR, Minton PA, Higgins SB, Hartert TV. Changes in urinary dinor dihydro F(2)-isoprostane metabolite concentrations, a marker of oxidative stress, during and following asthma exacerbations. Free Radic Res. 2007 Sep;41(9):956-62. doi: 10.1080/10715760701444600. PMID 17729112
- [Background] Britton JR, Pavord ID, Richards KA, Knox AJ, Wisniewski AF, Lewis SA, Tattersfield AE, Weiss ST. Dietary antioxidant vitamin intake and lung function in the general population. Am J Respir Crit Care Med. 1995 May;151(5):1383-7. doi: 10.1164/ajrccm.151.5.7735589.
- [Background] Fogarty A, Britton J. The role of diet in the aetiology of asthma. Clin Exp Allergy. 2000 May;30(5):615-27. doi: 10.1046/j.1365-2222.2000.00766.x. No abstract available. PMID 10792352
- [Background] Grievink L, Smit HA, Ocke MC, van 't Veer P, Kromhout D. Dietary intake of antioxidant (pro)-vitamins, respiratory symptoms and pulmonary function: the MORGEN study. Thorax. 1998 Mar;53(3):166-71. doi: 10.1136/thx.53.3.166. PMID 9659349
- [Background] Hatch GE. Asthma, inhaled oxidants, and dietary antioxidants. Am J Clin Nutr. 1995 Mar;61(3 Suppl):625S-630S. doi: 10.1093/ajcn/61.3.625S. PMID 7879729
- [Background] Miedema I, Feskens EJ, Heederik D, Kromhout D. Dietary determinants of long-term incidence of chronic nonspecific lung diseases. The Zutphen Study. Am J Epidemiol. 1993 Jul 1;138(1):37-45. doi: 10.1093/oxfordjournals.aje.a116775. PMID 8333425
- [Background] Comhair SA, Xu W, Ghosh S, Thunnissen FB, Almasan A, Calhoun WJ, Janocha AJ, Zheng L, Hazen SL, Erzurum SC. Superoxide dismutase inactivation in pathophysiology of asthmatic airway remodeling and reactivity. Am J Pathol. 2005 Mar;166(3):663-74. doi: 10.1016/S0002-9440(10)62288-2. PMID 15743779
- [Background] Comhair SA, Bhathena PR, Dweik RA, Kavuru M, Erzurum SC. Rapid loss of superoxide dismutase activity during antigen-induced asthmatic response. Lancet. 2000 Feb 19;355(9204):624. doi: 10.1016/S0140-6736(99)04736-4. PMID 10696986
- [Background] Gazak R, Walterova D, Kren V. Silybin and silymarin--new and emerging applications in medicine. Curr Med Chem. 2007;14(3):315-38. doi: 10.2174/092986707779941159. PMID 17305535
- [Background] Weyhenmeyer R, Mascher H, Birkmayer J. Study on dose-linearity of the pharmacokinetics of silibinin diastereomers using a new stereospecific assay. Int J Clin Pharmacol Ther Toxicol. 1992 Apr;30(4):134-8. PMID 1572758
- [Background] Wen Z, Dumas TE, Schrieber SJ, Hawke RL, Fried MW, Smith PC. Pharmacokinetics and metabolic profile of free, conjugated, and total silymarin flavonolignans in human plasma after oral administration of milk thistle extract. Drug Metab Dispos. 2008 Jan;36(1):65-72. doi: 10.1124/dmd.107.017566. Epub 2007 Oct 3. PMID 17913795
- [Background] Nelson SK, Bose SK, Grunwald GK, Myhill P, McCord JM. The induction of human superoxide dismutase and catalase in vivo: a fundamentally new approach to antioxidant therapy. Free Radic Biol Med. 2006 Jan 15;40(2):341-7. doi: 10.1016/j.freeradbiomed.2005.08.043. PMID 16413416
- [Background] Erzurum SC, Lemarchand P, Rosenfeld MA, Yoo JH, Crystal RG. Protection of human endothelial cells from oxidant injury by adenovirus-mediated transfer of the human catalase cDNA. Nucleic Acids Res. 1993 Apr 11;21(7):1607-12. doi: 10.1093/nar/21.7.1607. PMID 8479912
- [Background] Roberts LJ, Morrow JD. Measurement of F(2)-isoprostanes as an index of oxidative stress in vivo. Free Radic Biol Med. 2000 Feb 15;28(4):505-13. doi: 10.1016/s0891-5849(99)00264-6. PMID 10719231